CLINICAL TRIAL: NCT04405349
Title: A Multi-Centre, Open-label Phase 2a Trial of the Combination of VB10.16 and Atezolizumab in Patients With Advanced or Recurrent, Non-resectable HPV 16-Positive Cervical Cancer
Brief Title: Investigating the Combination of VB10.16 and Atezolizumab in Patients With HPV 16-positive Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nykode Therapeutics ASA (Industry)
Collaborators: Roche Pharma AG (Industry); Vaccibody AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB C-02
Record Dates: First submitted 2020-04-28; First posted 2020-05-28 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Cervical Cancer; Cervix Cancer
Keywords: Metastatic; Recurrent
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasm Metastasis; Recurrence | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental): VB10.16 vaccinations. 11 intramuscular (i.m.) vaccinations for up to 48 weeks from first vaccination. 5 vaccinations of 3 mg VB10.16 during the first 12 weeks, followed by vaccination every 6 weeks for up to 48 weeks + Atezolizumab (1200 mg) intravenous (i.v.) infusion every 3 weeks.
  Interventions: Biological: VB10.16; Biological: Atezolizumab

INTERVENTIONS:
Biological: VB10.16 — Vaccination
Biological: Atezolizumab — Intravenously infusion
  Other Names: Tecentriq

SUMMARY:
This phase IIa study is designed to evaluate the safety and efficacy of multiple dosing with VB10.16 immunotherapy in combination with atezolizumab in patients with advanced or recurrent non-resectable HPV16-positive cervical cancer, who failed or are not eligible for current standard of care.

DETAILED DESCRIPTION:
Patients will receive up to 11 intramuscular (i.m.) vaccinations of VB10.16, for up to 48 weeks from first vaccination. Patients will receive 5 vaccinations of 3 mg VB10.16 during the first 12 weeks, followed by vaccination every 6 weeks for up to 48 weeks from first immunisation (total of 11 vaccinations). Patients will receive up to 17 infusions of atezolizumab for up to 48 weeks from first treatment. Atezolizumab (1200 mg) will be administered as an intravenous (i.v.) infusion every 3 weeks. A follow-up period of up to 12 months will follow the 48 week treatment period.

Response to the VB10.16 and atezolizumab combination will be assessed by computed tomography (CT)/magnetic resonance imaging (MRI) at every 9 weeks throughout the treatment period according to the RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Has persistent, recurrent, or metastatic non-resectable squamous cell carcinoma, adeno-squamous carcinoma, or adenocarcinoma of the cervix, who has failed or is not eligible for treatment with systemic chemotherapy, radiotherapy or other standard-of-care anticancer treatment.
2. Tumour must be HPV16 positive. Provision of an archival tumour tissue sample not older than 2 years or new biopsy for analysing HPV16 status is mandatory.
3. Must have a biopsy (archived or new) available for PD L1 assessment at Screening.
4. Has measurable disease as assessed by the local site investigator/radiology as per RECIST 1.1.
5. Has recovered from the effects of surgery, radiation therapy, or chemoradiotherapy.
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1 at Screening.
7. Is aged 18 years or older.
8. Has life expectancy of at least 6 months in the best judgement of the investigator.
9. Is willing and able to sign a written informed consent form.

Exclusion Criteria:

1. Patients who, in the investigator's opinion, have progressed rapidly on their previous anticancer treatment (e.g., did not achieve any response [CR, PR, or SD]).
2. Has brain metastases (unless they have received prior treatment and are controlled and stable for at least 6 weeks before study enrolment) or leptomeningeal spread of disease.
3. Has positive serological test for hepatitis C virus (HCV), hepatitis B virus (HBV), surface antigen (HBsAg), positive HBV core antibody. Human immunodeficiency virus (HIV).
4. Has other concomitant or prior malignant disease,
5. Has an active, known or suspected autoimmune disease.
6. Is receiving systemic immunosuppression including systemic steroids or the use of immunosuppressive agents for any concurrent condition.
7. Has known allergy to aminoglycosides or kanamycin or any study treatment component.
8. Has history of toxic shock syndrome.
9. Has history of idiopathic pulmonary fibrosis, drug-induced pneumonitis, organising pneumonia, immune enteritis or active pneumonitis.
10. Has evidence or history of clinically significant cardiac disease including congestive heart failure
11. Has ongoing toxicity from prior therapy
12. Has severe infections within 4 weeks prior to study start
13. Current participation in a clinical trial
14. Has received investigational drug within 30 days before study entry.
15. Has received vaccination against infections within 30 days before study entry.
16. Has had prior treatment with CD137, anti-PD-1, or anti-PD-L1 therapeutic antibody or other immune checkpoint targeting agents.
17. Has known hypersensitivity to any component of the atezolizumab or VB10.16 formulation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | 48 weeks (1 year follow-up)
  The number and percentage of participants that experience an adverse event (AE
Overall response rate (ORR) using Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 at any time during the study | 48 weeks (1 year follow-up)
  ORR as assessed by RECIST v1.1

SECONDARY OUTCOMES:
Duration of response (DOR) | 48 weeks (1 year follow-up)
  Estimate the duration of response (DOR) in patients with advanced cervical cancer
Progression-free survival (PFS) | 48 weeks (1 year follow-up)
  Estimate the Progression-free survival (PFS) in patients with advanced cervical cancer
Overall survival (OS) | 48 weeks (1 year follow-up)
  Overall survival (OS) in patients with advanced cervical cancer
Evaluate immunogenicity of VB10.16 in combination with atezolizumab by analysing HPV16 E6/E7-specific cellular immune responses | 48 weeks (1 year follow-up)
  Systemic T-cell response

OTHER OUTCOMES:
Assess predictive biomarkers, such as programmed death-ligand 1 (PD-L1) in tumour material and investigate changes in tumour microenvironment by immunohistochemistry (IHC) and/or gene expression | 48 weeks (1 year follow-up)
  T cell infiltration, PD-L1 expression or other immune-oncology related genes
Correlating HPV16 circulating tumour DNA (ctDNA) in plasma with clinical response using RECIST 1.1 | 48 weeks (1 year follow-up)
  ctDNA

CONTACTS AND LOCATIONS:
Overall Officials: Siri Torhaug, MD, Study Director — Nykode Therapeutics ASA
Locations (21):
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hopital de Libramont, Brussels
  - Universitair Ziekenhuis Gent (Uz Gent), Ghent
  - Chu Ucl Namur, Namur
- Bulgaria (4):
  - Multiprofile Hospital for Active Treatment for Women's Health - Nadezhda Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment "Sv. Ivan Rilski", Sofia
  - Multiprofile Hospital for Active Treatment "Serdika"" EOOD, Sofia
  - University Multiprofile Hospital For Active Treatment Sofiamed, Sofia
- Czechia (4):
  - Masaryk Memorial Cancer Institute, Brno
  - Nemocnice Pardubickeho Kraje Pardubicka Nemocnice, Pardubice
  - University Hospital Kralovske Vinohrady, Prague
  - Nemocnice Na Bulovce, Prague
- Germany (5):
  - Universitatsklinikum Augsburg, Augsburg
  - University Clinic Carl Gustav Carus, Dresden
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Fakulat Mannheim Der Universitat Heidelberg, Heidelberg
- Oslo University Hospital, Oslo, Norway
- Poland (3):
  - Jagielońskie Centum Innowacji, Centrum Badań Klinicznych JCI, Krakow
  - Wielkopolskie Centrum Onkologii, Poznan
  - 'Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie, Warsaw

IPD SHARING:
Plan to Share IPD: No